CLINICAL TRIAL: NCT04808271
Title: The Effects of Bifidobacterium Breve Bif195 for Diarrhea-predominant Irritable Bowel Syndrome: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: The Effects of Bifidobacterium Breve Bif195 for Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Chr Hansen (Industry)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Principal Investigator, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-20060730
Record Dates: First submitted 2021-03-04; First posted 2021-03-22 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bif195 capsules (Active Comparator): The capsule will contain approximately 15*10^9 CFU of Bif195 per day. Excipients: Microcrystalline Cellulose 6 mg per capsule, Magnesium Stearate 1.5 mg per capsule, Maltodextrin 277.8 mg per capsule, and Sodium Ascorbate 14.7 mg per capsule.
  Interventions: Dietary Supplement: Bifidobacterium breve Bif195
- Placebo capsules (Placebo Comparator): The capsule contain only excipients: Microcrystalline Cellulose 6 mg per capsule, Magnesium Stearate 1.5 mg per capsule, Maltodextrin 277.8 mg per capsule, and Sodium Ascorbate 14.7 mg per capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium breve Bif195 — 1 capsule daily for 8 weeks
  Arms: Bif195 capsules
Dietary Supplement: Placebo — 1 capsule daily for 8 weeks
  Arms: Placebo capsules

SUMMARY:
The purpose of this study is to investigate if the probiotic Bifidobacterium breve Bif195 (Bif195) will result in improvement in clinical outcome in patients with diarrhea-predominant irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
IBS is the most frequently diagnosed gastrointestinal disease and also the most common cause of referrals to gastroenterology departments in Denmark.

The possibilities for treatment for IBS are limited. Treatment strategies that involve the microbiota provide symptom relief in some IBS patients. Several studies have demonstrated that the composition of the gut microbiota in IBS patients is different from healthy controls.

Probiotic interventions has shown promising results, but it currently remains unknown which probiotics are effective and which are not.

A new probiotic bacterium, Bifidobacterium breve Bif195 (Bif195) has been identified and has shown great effects on preventing enteropathy and ulcers on the gut mucosa in healthy volunteers given acetylsalicylic acid, and thereby Bif195 has also shown a potential in reducing gut permeability defects. This bacterium has not yet been investigated in IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IBS-D defined as more than one-fourth (25%) of bowel movements with Bristol Stool Scale Types 6-7 and less than one-fourth (25%) with Types 1-2
* Fulfill Rome IV diagnostic criteria for IBS
* Moderate to severe disease activity (IBS-SSS ≥175)
* Able to read and speak Danish
* Normal colonoscopy (performed within 1 year) if the patient had blood in stool

Exclusion Criteria:

* Other chronic gastro intestinal diseases including lactose intolerance and coeliac disease
* Fecal calprotectin ≥50 mg/kg
* Fecal sample positive for enteropathogenic microorganisms
* Surgical interventions in the GI region (except for appendectomy, hernia repair, cholecystectomy and gynecological and urological procedures)
* Psychiatric disorder
* Abuse of alcohol or drugs
* Medications except birth control pills, hormone supplements, allergies/asthma agents, blood pressure and cholesterol-lowering agents, proton pump inhibitors and non-prescription medicines; abnormal colonoscopy findings
* Pregnancy, planned pregnancy or breastfeeding females
* Ingestion of probiotics or antibiotics <4 weeks before the inclusion
* Abnormal screening biochemistry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Change in IBS symptoms from baseline measured by IBS-severity scoring system (IBS-SSS) at 8 weeks | 8 weeks
  IBS-SSS is a composite score of abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life. Each measure is rated from 0 to 100, with total scores ranging from 0 (best) to 500 (worst).

SECONDARY OUTCOMES:
Change in quality of life from baseline measured by Irritable Bowel Syndrome-Quality of Life (IBS-QOL) Questionnaire Scores at 8 weeks | 8 weeks
  The IBS-QoL questionnaire consists of 34 items, each with a 5-point response scale. The 34 items are based on the following eight variables: health worries, food avoidance, body image, dysphoria, interference with activity, social reactions, sexual activity and relationships. The IBS-QoL score will be transformed into a 0-100 scale using the formula: total score = (sum of the items-34/170) ×100. Low score (best)
Changes from baseline in bowel habits at 8 weeks | 8 weeks
  measured by frequency/day and Bristol Stool Form Scale. The Bristol Stool Form Scale is divided into seven categories were a low value indicate constipation and a high value indicate diarrhoea.
Change from baseline in abdominal pain at 8 weeks | 8 weeks
  Measured by a VAS scale from 0-10. 0 = no pain, 10 = worst pain
Adverse events | 16 weeks
  Reported according to IHC-GCP

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Copenhagen University, Hvidovre, Copenhagen
  - Copenhagen University Hospital Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gronbaek IMB, Halkjaer SI, Hansen EH, Mollerup S, Paulsen SJ, Konrad CV, Engel S, Bulinska-Balas M, Wellejus A, Haaber AB, Christensen AH, Engsbro AL, Petersen AM. Eight weeks of treatment with probiotic Bifidobacterium breve, Bif195 lowers fatigue scores in patients with diarrhoea-predominant irritable bowel syndrome: results from a randomised, clinical trial. Front Nutr. 2026 Jan 21;12:1701341. doi: 10.3389/fnut.2025.1701341. eCollection 2025. PMID 41648756